CLINICAL TRIAL: NCT03884361
Title: Does Elective Amniocentesis Change Vaginal Microbiome?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0126-18-HYMC
Record Dates: First submitted 2019-03-20; First posted 2019-03-21 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Vaginal Microbiome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaginal Microbiome as result of aminocentesis (Experimental): aginal Microbiome as result of aminocentesis by a blood and a vaginal samples that will taken before and after the aminocentesis
  Interventions: Diagnostic Test: Vaginal Microbiome as result of aminocentesis

INTERVENTIONS:
Diagnostic Test: Vaginal Microbiome as result of aminocentesis — we will take a blood samples and a vaginale samples after and before the aminicentesis and check if the sample that we took after is different and contain microrganisms , if we find a different o we can say that as result of the Elective Amniocentesis

SUMMARY:
the aim of this study is to check if elective amniocentesis change vaginal microbiome

ELIGIBILITY:
Inclusion Criteria:

* pregnant women between 18-45 years old , pregnant week is 16-24 , and a signle pregnant.

Exclusion Criteria:

* infection in the Uterus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-24 (Estimated); Study Completion 2021-03-24 (Estimated)

PRIMARY OUTCOMES:
Vaginal Microbiome | 1 year
  through blood and vaginal samples we will check if there are a vaginale micobiome - the samples will collected after and before the elective aminocentesis , the samples will sent to the labour of dr. Omer in the university , it will be analaysed there

CONTACTS AND LOCATIONS:
Overall Officials: Gabbay Gabbay Ben-Ziv, MD, Principal Investigator — Hillel Yaffe medical center, Hadera, Israel
Locations (1):
- Hillel Yaffe medical center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No